CLINICAL TRIAL: NCT00490594
Title: A Multi-Center Open Study to Evaluate the SeriACL™ Device for Primary Anterior Cruciate Ligament Repair
Brief Title: SeriACL™ Device Trial for Anterior Cruciate Ligament (ACL) Reconstruction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Serica Technologies, Inc. (Industry)
Responsible Party: Rebecca Horan, Serica Technologies, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-ACL1
Record Dates: First submitted 2007-06-20; First posted 2007-06-22 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Anterior Cruciate Ligament; Knee Injuries
Keywords: ACL; ligament; ACL injury
MeSH Terms: conditions — Knee Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ACL Reconstruction (SeriACL™ Device) — Bioresorbable ACL

SUMMARY:
The SeriACL device was developed as an alternative to an autograft (i.e., tissue that is taken from a patient's own body) or an allograft (i.e., tissue that is taken from a cadaver) for ACL reconstruction. The SeriACL device is made of silk yarns, knit and processed with SeriCoat™ surface treatment which makes it easier to wet the material. The SeriACL device is designed to be a temporary support structure to replace the torn ACL and to stabilize the knee joint following surgical repair. It is designed to use the body's own healing process to regenerate the patient's own new ligament tissue. As the new tissue grows and the support structure is needed less over time, the SeriACL device is bioresorbed (i.e., broken down) by the patient's body. The SeriACL device is designed to be installed with standard surgical techniques for ACL repair.

This study is designed to test the safety of the SeriACL device in primary total ACL repair in patients with a torn ACL. The study will evaluate whether repair of the ACL with the SeriACL device will return the knee to normal function and what, if any, side effects will occur.

ELIGIBILITY:
Inclusion Criteria:

* Complete ACL rupture
* Injured knee range of motion >= 75% of contralateral knee
* MCL tear grading <= 2
* Sign informed consent.

Exclusion criteria:

* Prior ACL reconstruction
* Complete PCL tear
* Locked bucket handle tear or complex tears of the menisci.
* Contralateral knee ligament injury
* Known joint disease
* Known allergy to silk
* Active drug or alcohol abuse
* Pregnant

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-06; Primary Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Safety - measured by device related SAEs | 12 months
KT-1000 Arthrometer | 12 months

SECONDARY OUTCOMES:
Knee Surveys | 12 months
Return to Work | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lars Engebretsen, MD, Principal Investigator — Ullevaal Hospital; Hans Paessler, MD, Principal Investigator — ATOS Clinic, Heidelberg; Holger Schmitt, MD, Principal Investigator — Heidelberg University
Locations (3):
- Germany (2):
  - Atos Clinic, Heidelberg
  - Heidelberg University, Heidelberg
- Ullevaal Hospital, Oslo, Norway